CLINICAL TRIAL: NCT00000656
Title: A Phase I/II, Open Label Study to Evaluate the Antiviral Potential of Combination Zidovudine and 2' 3'-Dideoxyinosine (Didanosine) in Patients With Asymptomatic HIV Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 143; 11118 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To assess the safety and to evaluate the anti-HIV effect of low-, moderate-, and high-dose schedules of zidovudine (AZT) plus didanosine (ddI) versus ddI alone in asymptomatic HIV-infected patients. Because of the failure with long-term (more than 1 year) use of, frequency of toxicity from, and drug resistance to AZT, drug combinations need to be developed to enable lower, less toxic doses of AZT to be used and to slow or prevent the development of resistance, while providing at least the same effectiveness.

DETAILED DESCRIPTION:
Because of the failure with long-term (more than 1 year) use of, frequency of toxicity from, and drug resistance to AZT, drug combinations need to be developed to enable lower, less toxic doses of AZT to be used and to slow or prevent the development of resistance, while providing at least the same effectiveness.

Enrollment during the first 8 weeks of the study is restricted to hemophiliacs and sexual partners of hemophiliacs with asymptomatic HIV disease. After the initial 8 weeks this restriction is lifted. Patients are randomized to one of four treatment arms with dosing of AZT plus ddI or ddI alone.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine.
* Acute and intermittent therapy with mycostatin and mycelex.
* Isoniazid, if no alternative therapy is available.

Allowed for up to 2 weeks:

* Acyclovir for Herpes infection (withhold didanosine during therapy).
* Acute therapy with fluconazole or ketoconazole.

Allowed but preferably not on a continuous basis for > 72 hours:

* Acetaminophen.
* Ibuprofen.
* Nonsteroidal antiinflammatory agents.

Patients must be:

* HIV antibody positive.
* Asymptomatic or have persistent generalized lymphadenopathy.
* Diagnosed with one of the listed coagulopathies.
* OR Sexual partner of someone with the above criteria.

Allowed:

* Basal cell carcinoma or in situ carcinoma of the cervix.

NOTE:

* As of January, 1991 full accrual of patients with prior AZT use has been reached - NOW ACCRUING ONLY THOSE WITH NO PRIOR AZT USE. Hemophilia restriction has been lifted.

Prior Medication:

Allowed:

* Zidovudine (AZT) for a total of = or < 13 months.

NOTE:

* As of January, 1991 accrual of these patients was reached, NOW ONLY PATIENTS WITH NO PRIOR AZT.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Unexplained temperature > 38 degrees C for more than 5 consecutive days or on more than 10 days in any 30-day period in the 2 years prior to study entry.
* Unexplained diarrhea defined as at least 3 liquid stools/day persisting more than 7 days within 2 years prior to study entry.
* Unintentional weight loss of > 10 pounds or > 10 percent of usual body weight within 2 years prior to study entry.
* Oral hairy leukoplakia at any time prior to study entry.
* Recurrent oral candidiasis unrelated to the use of antibiotics within 2 years prior to entry or unrelated to the use of antibiotics within the past 3 months.
* Herpes zoster within 2 years prior to study entry.
* Seizures within the past 6 months or currently requiring anticonvulsants for control.
* Current heart disease.
* Current psychological or emotional problems sufficient in the investigator's opinion to prevent adequate compliance with study therapy.
* Gout.

Concurrent Medication:

Excluded:

* Rifampin.
* Chemoprophylaxis for Pneumocystis carinii pneumonia other than aerosolized pentamidine.
* Intravenous pentamidine.
* Other antiretroviral agents, experimental medication, biological response modifiers, systemic corticosteroids, cimetidine, and ranitidine.
* Barbiturates.
* Oral acidifying agents.

Patients with a history of any of the following are excluded:

* AIDS-defining opportunistic infection, advanced AIDS-related complex, or malignancy.
* Acute or chronic pancreatitis.
* Grade 2 or higher neuropathy based on the Neuropathy Targeted Symptom Questionnaire.
* Seizures.
* Zidovudine therapy for = or > 13 months.
* Heart disease.
* Psychological or emotional problems sufficient in the investigator's opinion to prevent adequate compliance with study therapy.
* Gout.

Prior Medication:

Excluded within 4 weeks of study entry:

* Antiretroviral agents, including ribavirin, HPA-23, rifampin, AL721.
* Excluded within 3 months of study entry:
* Significant course of immunomodulating agents, such as steroids (> 1 week), isoprinosine, thymic factors, or any other experimental drugs.
* Excluded within 30 days prior to study entry:
* Neurotoxic drugs.

Excluded:

* Didanosine (ddI).
* Dideoxycytidine (ddC).
* Zidovudine (AZT) if received for > 13 months.

Prior Treatment:

Excluded within 3 months of entry:

* Other experimental therapy.

History of recent alcohol abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116
Dates: Study Completion 1993-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ragni MV, Study Chair; Merigan TC, Study Chair
Locations (5):
- United States (5):
  - Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California
  - Whitman - Walker Clinic, Washington D.C., District of Columbia
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Ragni MV, Amato DA, LoFaro ML, DeGruttola V, Van Der Horst C, Eyster ME, Kessler CM, Gjerset GF, Ho M, Parenti DM, et al. Randomized study of didanosine monotherapy and combination therapy with zidovudine in hemophilic and nonhemophilic subjects with asymptomatic human immunodeficiency virus-1 infection. AIDS Clinical Trial Groups. Blood. 1995 May 1;85(9):2337-46. PMID 7727768
- [Background] Mamtora G, Winters M, Drenkow J, Shafer R, Shen N, Tran H, Merigan T, Gingeras T. HIV-1 GeneChip and dideoxynucleotide sequence analysis of HIV-1 genomes present in plasma samples from patients of ACTG 143 study. Int Conf AIDS. 1996 Jul 7-12;11(1):221 (abstract no TuA265)
- [Background] Morse GD, Shelton MJ, Ho M, Bartos L, DeRemer M, Ragni M. Pharmacokinetics of zidovudine and didanosine during combination therapy. Antiviral Res. 1995 Aug;27(4):419-24. doi: 10.1016/0166-3542(95)00032-h. PMID 8540760
- [Background] Kozal M, Winters M, Shafer R, Kroodsma K, Katzenstein D, Merigan T. Behavior of codon 74 and 215 pol gene mutations in 62 AZT experienced patients on ddI monotherapy. Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:55
- [Background] Fiscus SA, DeGruttola V, Gupta P, Katzenstein DA, Meyer WA 3rd, LoFaro ML, Katzman M, Ragni MV, Reichelderfer PS, Coombs RW. Human immunodeficiency virus type 1 quantitative cell microculture as a measure of antiviral efficacy in a multicenter clinical trial. J Infect Dis. 1995 Feb;171(2):305-11. doi: 10.1093/infdis/171.2.305. PMID 7844365
- [Background] Winters MA, Shafer RW, Jellinger RA, Mamtora G, Gingeras T, Merigan TC. Human immunodeficiency virus type 1 reverse transcriptase genotype and drug susceptibility changes in infected individuals receiving dideoxyinosine monotherapy for 1 to 2 years. Antimicrob Agents Chemother. 1997 Apr;41(4):757-62. doi: 10.1128/AAC.41.4.757. PMID 9087484
- [Background] Shafer RW, Iversen AK, Kozal MJ, Winters MA, Katzenstein DA, Merigan TC. HIV-1 (HIV) isolates resistant to both AZT and ddI developing in patients receiving combination therapy contain unique pol gene mutations. Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:137
- [Background] Holodniy M, Katzenstein D, Winters M, Montoya J, Shafer R, Kozal M, Ragni M, Merigan TC. Measurement of HIV virus load and genotypic resistance by gene amplification in asymptomatic subjects treated with combination therapy. J Acquir Immune Defic Syndr (1988). 1993 Apr;6(4):366-9. PMID 8095981
- [Background] Shafer RW, Kozal MJ, Winters MA, Katzenstein DA, Ragni MV, Merigan TC. Combination therapy with ZDV+ddI suppresses virus load but does not prevent the emergence of HIV-1 isolates with ZDV resistance. ACTG 143 Protocol Virologists. Int Conf AIDS. 1993 Jun 6-11;9(1):68 (abstract no WS-B25-3)